CLINICAL TRIAL: NCT05603546
Title: A Prospective, Multicenter, Observational Study on the Treatment of Chronic Common Femoral Artery Bifurcation Occlusion
Acronym: EAST-CFA
Status: Recruiting | Type: Observational
Sponsor: Qingdao Hiser Medical Group (Other)
Responsible Party: Sponsor
Other Study IDs: the EAST-CFA study
Record Dates: First submitted 2022-02-13; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-01

CONDITIONS: Common Femoral Artery Occlusive Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CFA treated by endarterectomy: Common femoral artery lesions undergo endometrial decortication
- CFA treated by transluminal extraction-atherectomy: Common femoral artery lesions are treated intravenously

SUMMARY:
This study is a prospective, multicenter real-world observational study to understand the safety and efficacy of endoluminal therapy and traditional endometristomy in the real world for patients with severe stenosis and occlusion of the common femoral artery. The study will enroll 300 patients with severe stenosis and occlusion of chronic common femoral artery in nine centers across the country. According to the different intervention methods of the common femoral artery, the enrolled cases were divided into two groups: A: endometrial detachment for common femoral artery lesions and B: interventional endovascular treatment for common femoral artery lesions. As it is a real-world study, there is no separate primary endpoint indicator, which mainly observes F-TLR (immunity from vascular re-intervention), technical success rate, duration of surgery, length of hospital stay, common femoral artery patency rate, deep femoral artery patency rate, direct and indirect medical expenditure associated with the disease in 24 months, MAE (major adverse events), and perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic atherosclerotic occlusion who are over 18 years old;
2. Patients with Rutherford clinical grading range in the range of 2-5;
3. The stenosis rate of the common femoral artery (including the bifurcation of the femoral artery) is > 60% or occlusive, and it is proposed to undergo intraluminal treatment such as balloon dilation, stent implantation, plaque rotation and excision, or endometrial decortication treatment;
4. At least one healthy sub-knee outflow tract (or opened through reconstruction) communicates with the blood vessels of the foot;
5. Intravascular treatment: the guide wire successfully passed through the target lesion;
6. For patients with combined aorta iliac artery lesions, after completing the reconstruction of the main iliac artery, they can be enrolled according to the above requirements; except for the ipsilateral iliac artery, other non-target lesions of the remaining non-target blood vessels can be treated by the doctor at his own discretion;
7. For patients with both lower limbs that meet the admission conditions, both limbs can be enrolled separately in chronological order;
8. Written informed consent prior to the study procedure.

Exclusion Criteria:

1. Patients who are unwilling or refuse to sign informed consent;
2. Known or suspected allergy or contraindications to aspirin, clopidogrel bisulfate, heparin or contrast agents;
3. Patients who have participated in clinical trials of other drugs or medical devices that interfere with this clinical trial in the past 3 onths;
4. pregnant and lactating women;
5. Life expectancy is less than 24 months;
6. Patients whose common femoral artery has received endometrial detachment, plaque rotation, stent implantation and restenosis in stents;
7. Patients with acute ischemia of grade III lower extremities who have lost the opportunity for vascular reconstruction;
8. Any major medical condition that the researchers believe may affect the subject's optimal participation in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with severe chronic primary stenosis or occlusion of the common femoral artery (including the femoral artery bifurcation) requiring endovascular therapy or plaque stripping were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-02-14 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
Major adverse events | post-interventional 30days
  Major adverse events at 30days
freedom from target lesion revascularization | post-interventional 2 years
  freedom from target lesion revascularization at 2years

SECONDARY OUTCOMES:
Technical success rate | post-intervention
Time of surgery | post-intervention
Time of hospital stay | post-hospitalization
primary patency of CFA | post-interventional 1,3,6, 9,12 and 24 month
  primary patency of CFA at 1,3,6, 9,12 and 24 month
primary patency of PFA | post-interventional 1,3,6, 9,12 and 24 month
  primary patency of CFA at 1,3,6, 9,12 and 24 month
freedom from target lesion revascularization | post-interventional 1,3,6, 9,12 month
  freedom from target lesion revascularization at 1,3,6, 9,12 month
Perioperative complications | post-interventional 30days
  Perioperative complications at 30days
Direct and indirect medical expenditures associated with the disease | post-hospitalization 24 months
  Direct and indirect medical expenditures associated with the disease at 24months

CONTACTS AND LOCATIONS:
Locations (1):
- Hiser Medical Group, Qingdao, Shandong, China